CLINICAL TRIAL: NCT04509245
Title: The Effects of a Novel Real Food Based Digital Education-assisted Lifestyle Intervention Program on Metabolism in Type 2 Diabetes
Brief Title: The Effects of a Novel Lifestyle Intervention Program on Insulin Sensitivity in Type 2 Diabetes
Acronym: CH_DDZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Changing_Health_DDZ
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes; Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effects of a digitally assisted lifestyle intervention (Experimental): Testing the effects of a low-calorie diet in connection with app-based digital education and behavioral change program on glucose metabolism and disease management.
  Interventions: Behavioral: Low-calorie diet supported by an app-guided digital education program, nutritional coaching calls via phone

INTERVENTIONS:
Behavioral: Low-calorie diet supported by an app-guided digital education program, nutritional coaching calls via phone — During the 12-week intervention participants were asked to adhere to a real food-based low-calorie diet supported by an app-guided digital education program as well as a low-calorie recipe book and received weekly coaching calls by nutritionists

SUMMARY:
Moderate weight reduction by a moderately hypocaloric very-low-fat diet resulted in normalization of fasting hyperglycemia and reversal of hepatic insulin resistance in patients with poorly controlled type 2 diabetes. The Diabetes Remission Clinical Trial (DiRECT) revealed that utilizing a total diet replacement by a low-energy formula diet for 3 months led to a 15 kg or more weight loss in 24% participants and diabetes remission 46% of the participants. To date it remains unknown whether similar results can be achieved with a natural, non-formula based diet in connection with an educative smartphone application and telephone coaching

DETAILED DESCRIPTION:
24 patients with type 2 diabetes from the German Diabetes Study (GDS) with less than 4 years disease duration and not receiving insulin were included in this study. Before the start of the intervention, participants documented their dietary intake by recording a food diary. During the 12-week intervention participants were asked to adhere to a real food-based low-calorie diet supported by an app-guided digital education program as well as a low-calorie recipe book and received weekly coaching calls by nutritionists. Patients were instructed to adhere to a balanced low calorie diet during the intervention. Nutritionists provided structured behavior change focusing on dietary advice, adherence to logging dietary intake and tracking weight. At first visit, patients installed the Changing Health App (Changing Health, Newcastle, UK) and completed an app-based digital education program. This program focused on type 2 diabetes education and behavioral change in combination with weight tracking and dietary monitoring. Patients used the app throughout the study and adherence was monitored via logins. Comprehensive testing before and after the intervention comprised a mixed-meal tolerance test and liver fat.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Existing diagnosis of type 2 diabetes
* Individuals who use a smartphone or PC to install the app
* Individuals who are able to communicate in German

Exclusion Criteria:

* Physical disability that leads to a significant lack of mobility (wheelchair, walking aid, walking stick, cane or crutches)
* Insulin therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Change in insulin sensitivity after 12 weeks of intervention
  Change in insulin sensitivity can be estimated via a mixed-meal tolerance test, a standardized liquid meal consumed by the participants

SECONDARY OUTCOMES:
Change in öiver fat | Change in liver fat after 12 weeks of intervention
  Change in liver fat content was estimated from 1-Proton-Magnetic Resonance Spectroscopy in a human scanner

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, MD, Principal Investigator — German Diabetes Center
Locations (1):
- DDZ (Deutsches Diabetes Zentrum), Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaharia OP, Kupriyanova Y, Karusheva Y, Markgraf DF, Kantartzis K, Birkenfeld AL, Trenell M, Sahasranaman A, Cheyette C, Kossler T, Bodis K, Burkart V, Hwang JH, Roden M, Szendroedi J, Pesta DH. Improving insulin sensitivity, liver steatosis and fibrosis in type 2 diabetes by a food-based digital education-assisted lifestyle intervention program: a feasibility study. Eur J Nutr. 2021 Oct;60(7):3811-3818. doi: 10.1007/s00394-021-02521-3. Epub 2021 Apr 11. PMID 33839905